CLINICAL TRIAL: NCT04071977
Title: Effect of Combined Antioxidant Therapy on the Levels of Oxidative Stress Markers in Aqueous and Vitreous Humor of Patients With Proliferative Diabetic Retinopathy
Brief Title: Combined Antioxidant Therapy on Oxidative Stress in Aqueous and Vitreous Humor of Diabetic Retinopathy Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Guadalajara (Other)
Collaborators: Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, Adolfo Daniel Rodriguez-Carrizalez, Clinical Professor, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RD-20180831
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Diabetic Retinopathy; Oxidative Stress; Diabetes
Keywords: Vitreous humor; Vitrectomy; Aqueous humor; Antioxidant therapy; Oxidative markers
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus | interventions — Magnesium Oxide

STUDY DESIGN:
Intervention Model Description: Clinical trial phase IIa
Who Masked: Participant, Investigator
Masking Description: Drug
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined Antioxidant Therapy group (Active Comparator): This arm will be administered with the combined antioxidant therapy, and will consist of 28 patients with proliferative diabetic retinopathy (PDR) who will undergo vitrectomy.
  Interventions: Drug: Combined antioxidant therapy
- Placebo group (Placebo Comparator): This arm will be administered with placebo, and will consist of 28 patients with proliferative diabetic retinopathy (PDR) who will undergo vitrectomy.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Combined antioxidant therapy — It consists of a tablet with lutein (10 mg), astaxanthin (4 mg), Zeaxanthin (1 mg), vitamin C (L-ascorbic acid 180 mg), vitamin E (DL-alpha tocopherol 30 mg), zinc (zinc oxide 20 mg), copper (copper sulfate 1 mg), taken once a day for 12 months
  Other Names: Drusen Laz
  Arms: Combined Antioxidant Therapy group
Other: Placebo — It consists in a capsule with 100 mg of magnesium oxide
  Other Names: Magnesia
  Arms: Placebo group

SUMMARY:
The present study aims to support previous research on the effects of antioxidant therapy on the outcome of diabetic retinopathy and local oxidative stress values. The researchers intend to evaluate 56 patients with proliferative diabetic retinopathy undergoing the vitrectomy procedure, who will be assigned to a placebo group or combination antioxidant therapy. Each group will receive the intervention for 2 months. This intervention consists of taking one tablet (placebo or antioxidant therapy) orally, once a day.

At the beginning of the study, only blood samples will be collected to evaluate the state of oxidative and metabolic stress at a systemic level. After 2 months of intervention, blood samples will be taken again on the day of the intervention, adding the samples of aqueous and vitreous humor obtained during the vitrectomy. The results obtained between both groups and the different analysis matrices will be compared.

DETAILED DESCRIPTION:
Diabetic retinopathy is a diabetes microvascular complication due to an insufficient oxygen supply to its endothelial cells in states of constant hyperglycemia. This entity is classified in two main categories: non-proliferative diabetic retinopathy and proliferative diabetic retinopathy, the latter is characterized for the presence of neovascularization as oppose to the first one.

Oxidative stress has been considered as one of the main factors in the development of diabetic retinopathy. It is a result from an imbalance between oxidants production and cellular antioxidant defenses, which provokes DNA damage.

The treatment of diabetic retinopathy simply includes glycemic, lipemic and blood pressure control. Only when the view is compromised is when a vitrectomy is performed, which usually occurs in the more advanced stages such as the proliferative stage. Antioxidant therapy has been used as a coadjuvant for these interventions, complementing the action and efficacy of the treatment established for diabetic retinopathy in the early stages. However, in order to obtain vitreous and aqueous humor, the vitrectomy procedure is required, which is only carried out in the proliferative stage.

Diabetic retinopathy is a specific and chronic complication of diabetes mellitus and is known to have a prevalence of 43.6% internationally and 31.5% in the Mexican population. It represents the main cause of visual blindness and weakness in the economically active population, which also affects the quality of life and the productivity of the people who suffer it.

The researchers intend to evaluate whether antioxidant therapy influences the levels of oxidative stress markers at the ocular level.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 with proliferative diabetic retinopathy
* Blood pressure under 160/100 mmHg
* HbA1c equal or lower than 9%
* LDL under 190mg/dl, triglycerides under 500mg/dl)
* Signed informed consent
* Patients scheduled for vitrectomy surgery, under the following indications:
* Severe vitreous hemorrhage lasting 1-3 months or longer, which does not go away spontaneously
* Rhegmatogenous or tensile retina detachment
* Epiretinal membrane that involves macula and that includes vitreomacular traction

Exclusion Criteria:

* Vitreous hemorrhage for any cause other than Proliferative Diabetic Retinopathy complication
* Patients with vitrectomy surgery in the last 6 months
* Patients with laser surgery in the last 6 months
* Intravitreal application of antiangiogenic agents in the last 2 months
* Patients with other ocular pathologies such as age-related macular degeneration, glaucoma, endophthalmitis, conjunctivitis of any etiology, severe lacrimal film dysfunction syndrome, etc.
* Patients with concomitant systemic diseases such as: rheumatoid arthritis, sjogren's syndrome, upper respiratory tract infections, gastrointestinal infections, sepsis, any infectious process
* Patients with severe cardiovascular disease (myocardial infarction, stroke, severe peripheral vascular disease)
* Oral antioxidant intake that exceeds the daily recommendations in the last 6 months.
* Consumption of pharmacological agents such as: immunomodulators, biological, anti-inflammatory, in the last 3 months
* Smokers
* Patients with neurodegenerative or carcinogen processes
* Patients who are currently participating in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-03-25 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Compare levels of markers of oxidative stress in aqueous humor and vitreous humor | 1 measure will be made after 2 months of intervention
  The investigators will measure oxidative stress markers in aqueous and vitreous humor taken during vitrectomy procedure and compare such results between both intervention groups.
Changes in concentration of plasma 8-isoprostanes after intervention. | 2 measures will be made, 1 at baseline, and one after completion of 2 months of intervention
  The investigators will consider changes presented in plasma concentrations of 8-isoprostanes from baseline to the end of the intervention. The investigators expect to find a decrease in 8-isoprostanes concentrations in the supplemented group.
Changes in concentration of total antioxidant capacity (TAC) after intervention from baseline. | 2 measures will be made, 1 at baseline, and one after completion of 2 months of intervention
  The investigators will consider changes presented in plasma concentrations of total antioxidant capacity (TAC) from baseline to the end of the intervention. The investigators expect to find TAC augmentation in the supplemented group.

SECONDARY OUTCOMES:
Correlate the levels of 8-isoprostanes in systemic samples, aqueous humor and vitreous humor with the glycosylated hemoglobin value of patients with proliferative diabetic retinopathy. | 1 measure of glycated hemoglobin will be taken at baseline
  The investigators will consider levels of 8-isoprostanes in serum, aqueous humor and vitreous humor after intervention and baseline glycated hemoglobin
Correlate the levels of total antioxidant capacity (TAC) in systemic samples, aqueous humor and vitreous humor with the glycosylated hemoglobin value of patients with proliferative diabetic retinopathy. | 1 measure of glycated hemoglobin will be taken at baseline
  The investigators will consider levels of total antioxidant capacity in serum, aqueous humor and vitreous humor after intervention and baseline glycated hemoglobin

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Experimental and Clinical Therapeutics,, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rodriguez-Carrizalez AD, Castellanos-Gonzalez JA, Martinez-Romero EC, Miller-Arrevillaga G, Villa-Hernandez D, Hernandez-Godinez PP, Ortiz GG, Pacheco-Moises FP, Cardona-Munoz EG, Miranda-Diaz AG. Oxidants, antioxidants and mitochondrial function in non-proliferative diabetic retinopathy. J Diabetes. 2014 Mar;6(2):167-75. doi: 10.1111/1753-0407.12076. Epub 2013 Aug 21. PMID 23875878
- [Background] Rodriguez-Carrizalez AD, Castellanos-Gonzalez JA, Martinez-Romero EC, Miller-Arrevillaga G, Roman-Pintos LM, Pacheco-Moises FP, Miranda-Diaz AG. The antioxidant effect of ubiquinone and combined therapy on mitochondrial function in blood cells in non-proliferative diabetic retinopathy: A randomized, double-blind, phase IIa, placebo-controlled study. Redox Rep. 2016 Jul;21(4):190-5. doi: 10.1179/1351000215Y.0000000032. Epub 2016 Feb 5. PMID 26207797
- [Background] Rodriguez-Carrizalez AD, Castellanos-Gonzalez JA, Martinez-Romero EC, Miller-Arrevillaga G, Pacheco-Moises FP, Roman-Pintos LM, Miranda-Diaz AG. The effect of ubiquinone and combined antioxidant therapy on oxidative stress markers in non-proliferative diabetic retinopathy: A phase IIa, randomized, double-blind, and placebo-controlled study. Redox Rep. 2016 Jul;21(4):155-63. doi: 10.1179/1351000215Y.0000000040. Epub 2015 Aug 31. PMID 26321469
- [Background] Sonia Sifuentes-Franco, Adolfo Daniel Rodríguez-Carrizalez, Sandra Carrillo- Ibarra, José Alberto Castellanos-González, Esaú César Martínez-Romero, Guillermo Miller-Arrevillaga and Alejandra Guillermina Miranda-Díaz. The effect of Ubiquinone administration on oxidative DNA damage and repair in plasma levels in non-proliferative diabetic retinopathy.Diabetes Management 2017;7(2):186-191
- [Background] Cecilia OM, Jose Alberto CG, Jose NP, Ernesto German CM, Ana Karen LC, Luis Miguel RP, Ricardo Raul RR, Adolfo Daniel RC. Oxidative Stress as the Main Target in Diabetic Retinopathy Pathophysiology. J Diabetes Res. 2019 Aug 14;2019:8562408. doi: 10.1155/2019/8562408. eCollection 2019. PMID 31511825
- [Background] Robles-Rivera RR, Castellanos-Gonzalez JA, Olvera-Montano C, Flores-Martin RA, Lopez-Contreras AK, Arevalo-Simental DE, Cardona-Munoz EG, Roman-Pintos LM, Rodriguez-Carrizalez AD. Adjuvant Therapies in Diabetic Retinopathy as an Early Approach to Delay Its Progression: The Importance of Oxidative Stress and Inflammation. Oxid Med Cell Longev. 2020 Mar 11;2020:3096470. doi: 10.1155/2020/3096470. eCollection 2020. PMID 32256949
- [Background] Lopez-Contreras AK, Martinez-Ruiz MG, Olvera-Montano C, Robles-Rivera RR, Arevalo-Simental DE, Castellanos-Gonzalez JA, Hernandez-Chavez A, Huerta-Olvera SG, Cardona-Munoz EG, Rodriguez-Carrizalez AD. Importance of the Use of Oxidative Stress Biomarkers and Inflammatory Profile in Aqueous and Vitreous Humor in Diabetic Retinopathy. Antioxidants (Basel). 2020 Sep 20;9(9):891. doi: 10.3390/antiox9090891. PMID 32962301